CLINICAL TRIAL: NCT05596214
Title: Combination of Curcumin and Berberine Therapy in the Treatment of Post Acute Diverticulitis (AD) Symptomatic Uncomplicated Diverticular Disease (SUDD)
Brief Title: Combination of Curcumin and Berberine Therapy in the Treatment of Post Acute Diverticulitis (SUDD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Adi Lahat (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Adi Lahat, Principal Investigator, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7824-20-SMC
Record Dates: First submitted 2022-09-18; First posted 2022-10-27 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Diverticulitis
MeSH Terms: conditions — Diverticulitis | interventions — Coptis extract

STUDY DESIGN:
Intervention Model Description: 2 Stage study: Stage 1 will comprise an open label single arm exploratory study of 10 patients suffering from post AD SUDD investigating oral Cur-Berberine (Coptis) therapy for induction of clinical response.
  Stage 2: If clinical response is achieved in ≥ 3 patients and no significant safety signals will emerge, we will proceed to a prospective pilot randomized placebo-controlled study.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curcumin-Berberine (coptis) therapy (Experimental): Cur-Berberine (Coptis) treatment will consist: 2 capsules of 500 mg Berberine (Coptis) before breakfast (a total of 1.0gr Berberine) and 3 capsules of 500mg curcumin before dinner (a total of 1.5gr curcumin).
  Interventions: Combination Product: Curcumin-Berberine (coptis)
- Placebo (Placebo Comparator): 2 capsules of 500 mg placebo before breakfast and 3 capsules of 500mg placebo before dinner.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: Curcumin-Berberine (coptis) — dietary supplement
  Arms: Curcumin-Berberine (coptis) therapy
Combination Product: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Curcumin (Cur), an active ingredient of the Indian herb Rhizoma Curcuma Longa, has been extensively studied in the context of inflammatory diseases. Studies have demonstrated its efficacy in reducing chemically induced colitis in animal models and in humans.

Berberine is a phytochemical derived from plants such as coptis chinensis, goldenseal and scutellaria. These herbal remedies have been used in both Chinese and European medicine for centuries to treat digestive inflammation and infectious diseases.

Therefore the investigator see a possible dual mechanism of curcumin-Berberine (Coptis) treatment in SUDD patients through both direct anti-inflammatory action and modulation of intestinal microbiome.

This data provides basis for investigating an integrative approach to optimize and offer treatment to patients suffering from post AD SUDD. The investigator speculate that using a combined gut-directed formulation of curcumin-Berberine could benefit this subgroup of patients and improve their clinical symptoms.

DETAILED DESCRIPTION:
The objective of the study is to investigate the efficacy and safety of gut-directed enteric-coated curcumin-Berberine (Coptis) combination therapy to induce remission in patients suffering from post AD SUDD.

Methods:

This will be a two-stage study:

Stage 1 will comprise an open label single arm exploratory study of 10 patients suffering from post AD SUDD investigating oral Cur-Berberine (Coptis) therapy for induction of clinical response.

Stage 2: If clinical response is achieved in ≥ 3 patients and no significant safety signals will emerge, the investigator will proceed to a prospective pilot randomized placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of previous acute diverticulitis (AD) and on-going abdominal symptoms comprising a SUDD (left abdominal pain and/or change in bowel habits and bloating)
2. Having an active SUDD defined by Diverticular Clinical Score (DICS) score ≥10.
3. Age 18-80 years.
4. Able and willing to give written consent

   -

Exclusion Criteria:

1. Patient with non-controlled renal or liver disease, hypertension, cardiovascular disease, cerebrovascular disease, chronic pancreatitis, diabetes mellitus, gallstone disease, uncontrolled migraines or neurological disorders
2. Patients with significant laboratory abnormalities, including anemia with hemoglobin <10, leucopenia (WBC<4k/mcl), thrombocytopenia (Plt<100K/mcl), abnormal coagulation tests (INR, PTT), or elevation of liver or kidney function tests above the normal values.
3. Patient with active infection, sepsis or pneumonia.
4. Pregnant or nursing women.
5. Unable or unwilling to receive Curcumin-Berberine (Coptis) therapy
6. Known allergy to either curcumin or Berberine (Coptis)

   -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-14 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients reaching clinical response after initiation of therapy. | 8 weeks
  Clinical response is defined as a drop of ≥3 points of the DICS score.

SECONDARY OUTCOMES:
Percentage of patients who had a clinical remission after initiation of therapy. | 8 weeks
  Clinical remission is defined as DICS score ≤ 5 within 4 weeks.
Percentage of patients who had a rapid clinical response after induction of therapy. | 8 weeks
  Clinical response is defined as a drop of ≥3 points of the DICS score
Percentage of patients who achieve normalization and/or >50% improvement of CRP and/or calprotectin levels (computed out of patients with abnormal values at baseline for these indices). | 8 weeks
  Calculation of the percentage of patients who achieve improvement of CRP
Time-to-response defined as number of days to achieve a drop of ≥3 points of the DICS score. | 8 weeks
  Within how many days the patient achieved drop of points in the DICS questionnaire
The percentage of patients in clinical remission at day 7 after induction of therapy. | Within 7 days
  Calculation of the percentage of patients achieved clinical remission at day 7

CONTACTS AND LOCATIONS:
Overall Officials: Adi Lahat-Zok, MD, Principal Investigator — Gastroenterology department, Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No